CLINICAL TRIAL: NCT03699228
Title: China Nationwide Multi Center Big Data Study on the Quantitative Computed Tomography (QCT) and Health Status of Check -up Population
Brief Title: China Health Big Data
Acronym: China biobank
Status: Recruiting | Type: Observational
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other); Ruijin Hospital (Other); Huashan Hospital (Other); Henan Provincial People's Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The renmin hospital of wuhan university (Unknown); Nanjing BenQ Hospital (Unknown); China-Japan Friendship Hospital (Other); xinan hospital (Unknown); Wu Hu Yijishan hospital (Unknown); The fifth affiliated hospital of zhong shan university (Unknown)
Responsible Party: Principal Investigator, xiaoguang Cheng, professor of radiology, chairman of department, Beijing Jishuitan Hospital
Other Study IDs: jst2018
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-02

CONDITIONS: Osteoporosis; Obesity; Liver Steatoses
Keywords: Bone mineral density, quantitative computed tomography, Osteoporosis, obesity, liver steatosis
MeSH Terms: conditions — Osteoporosis; Obesity; Fatty Liver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this nationwide multi center study the investigators combine the low dose chest CT scan data with QCT technology, to measure the BMD of spine, VAT and liver fat in the health check subjects. The aim of this study is to evaluate the performance of QCT in the health check field, and further to evaluate the prevalence of osteoporosis, obesity and liver steatosis in health check population across China.

DETAILED DESCRIPTION:
Low dose Chest CT scan is the standard for lung cancer in the health check center in China. Quantitative computed tomography (QCT) is utilizing the CT raw data to measure the bone mineral density (BMD), the visceral fat (VAT) and liver fat content in human, which can be widely used in the diagnosis of osteoporosis, the assessment of obesity and liver steatosis. In this nationwide multi center study the investigators combine the low dose chest CT scan data with QCT technology, to measure the BMD of spine, VAT and liver fat in the health check subjects. This study is to evaluate the performance of QCT in the health check field, and further to evaluate the prevalence of osteoporosis, obesity and liver steatosis in health check population across China.

ELIGIBILITY:
Inclusion Criteria:

health check subjects 30-90 years old low dose chest CT scan

Exclusion Criteria:

pregnant women metal implant in the CT scan area

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General health check population
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The spinal volumetric bone mineral density (vBMD) | 2 year
  The volumetric bone mineral density of L1-2 measured by QCT

SECONDARY OUTCOMES:
The visceral adipose tissue (VAT) | 2 year
  The visceral adipose tissue (VAT) measured by quantitative computed tomography (QCT)
Liver fat | 2 years
  Liver fat measurement by quantitative computed tomography (QCT)

CONTACTS AND LOCATIONS:
Overall Officials: xiaoguang cheng, MD, Principal Investigator — Beijing Jishuitan Hospital; qiang zeng, Principal Investigator — General PLA hospital
Locations (6):
- China (6):
  - Wu Hu Yijishan Hospital, Wuhu, Anhui
  - Beijing Jishuitan hospital, Beijing, Beijing Municipality
  - The first affiliated hospital of Guiyang Medical University, Guiyang, Guizhou
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Hua Shan hospital, Shanghai, Shanghai Municipality
  - Shanghai Ruijin hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Sun Y, Qi X, Wang X, Lin X, Zhou Y, Du Y, Liu A, Lv X, Zhou J, Li Z, Wu X, Zou Z, Zhang M, Zhu J, Shang F, Li Y, Li H. Association between high-density lipoprotein cholesterol and lumbar bone mineral density in Chinese: a large cross-sectional study. Lipids Health Dis. 2024 Jan 24;23(1):27. doi: 10.1186/s12944-024-02023-1. PMID 38267987
- [Derived] Sun Y, Qi X, Lin X, Zhou Y, Lv X, Zhou J, Li Z, Wu X, Zou Z, Li Y, Li H. Association between total cholesterol and lumbar bone density in Chinese: a study of physical examination data from 2018 to 2023. Lipids Health Dis. 2023 Oct 21;22(1):180. doi: 10.1186/s12944-023-01946-5. PMID 37865752
- [Derived] Cheng X, Zhao K, Zha X, Du X, Li Y, Chen S, Wu Y, Li S, Lu Y, Zhang Y, Xiao X, Li Y, Ma X, Gong X, Chen W, Yang Y, Jiao J, Chen B, Lv Y, Gao J, Hong G, Pan Y, Yan Y, Qi H, Ran L, Zhai J, Wang L, Li K, Fu H, Wu J, Liu S, Blake GM, Pickhardt PJ, Ma Y, Fu X, Dong S, Zeng Q, Guo Z, Hind K, Engelke K, Tian W; China Health Big Data (China Biobank) project investigators. Opportunistic Screening Using Low-Dose CT and the Prevalence of Osteoporosis in China: A Nationwide, Multicenter Study. J Bone Miner Res. 2021 Mar;36(3):427-435. doi: 10.1002/jbmr.4187. Epub 2020 Nov 4. PMID 33145809